CLINICAL TRIAL: NCT01300598
Title: Safety and Efficacy of Autologous Adipose Tissue Derived Mesenchymal Stem Cells Transplantation in Patient With Degenerative Arthritis
Brief Title: Autologous Adipose Tissue Derived Mesenchymal Stem Cells Transplantation in Patient With Degenerative Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: R-Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Jointstem
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Degenerative Arthritis
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Procedure: Autologous Adipose Tissue derived MSCs Transplantation — Intra-articular infusion of Autologous Adipose Derived Mesenchymal Stem Cells. Dose : 1x10e7 cells/3mL,5x10e7 cells/3mL, 1x10e8 cells/3mL
  Other Names: RNL-JointStem®

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of autologous transplantation of Adipose Tissue derived Mesenchymal stem cells (MSCs) in patient with degenerative arthritis.

DETAILED DESCRIPTION:
degenerative arthritis is the most common type of arthritis. It is estimated that 26.9 million Americans 25 years old or older have clinical degenerative arthritis of some joints, with a higher percentage of affliction in the older population. Its clinical manifestations include joint pain and impairment to movement, and surrounding tissues are often affected with local inflammation. The etiology of degenerative arthritis is not completely understood; however, injury, age, and genetics have been considered among the risk factors.

Degenerative arthritis is a progressively debilitating disease that affects mostly cartilage, with associated changes in bone. Cartilage has limited intrinsic healing and regenerative capacities.

Due to the increasing incidence of degenerative arthritis and the aging population coupled with inefficient therapeutic choices, novel cartilage repair strategies are in need.

The availability of large quantities of MSCs and their potential for ready chondrogenic differentiation after prolonged in vitro expansion have made MSCs the most hopeful candidate progenitor cell source for cartilage tissue engineering.

In the clinical study, mesenchymal stem cells will be isolated from adipose tissue and cultured, and administered into the cartilage tissue lesion by orthopedic surgery.

It will be stimulate the regeneration of defective cartilage tissue and to improve their functions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who understand and sign the consent form for this study.
* Age :18-75, males and females.
* Clinical diagnosis of degenerative arthritis by Radiographic Criteria of Kellgren and Lawrence.
* Patients who can't treat with traditional medication and need a arthroplasty.
* Patients whose lesion is 2~6 cm2 in size.
* Duration of pain over Grade 4(11-point numeric scale) : > 4 months

Exclusion Criteria:

* Women who are pregnant or breast feeding or planning to become pregnant during the study.
* Objects who administer with a anti-inflammatory drugs contain herbal medicine within 14 days prior to inclusion in the study.
* History or current evidence of alcohol or drug abuse or is a recreational user of illicit drugs or prescription medications.
* Treatment with intra-articular injection therapy within 2 months prior to screen.
* Other joint diseases except degenerative arthritis : systemic or rheumatic or inflammatory chondropathy, chondrocalcinosis, hemachromatosis, inflammatory joint disease, avascular necrosis of the femoral head, Paget's disease, hemophilic arthropathy, infectional arthritis, Charcot's disease, villonodular synovitis, synovial chondromatosis.
* Positive serology for HIV-1 orHIV-2, Hepatitis B (HBsAg, Anti-HCV-Ab), Hepatitis C (Anti-HCV-Ab) and syphilis.
* Serious pre-existing medical conditions like Cardiovascular Diseases, Renal Diseases, Liver Diseases, Endocrine Diseases, Cancer and Diabetes Mellitus.
* Overweight expressed as body mass index (BMI) greater than 30 (obesity grade II). BMI estimated as mass (kg) / corporal surface (m2).
* Participation in another clinical trial or treatment with a different investigational product within 3 months prior to inclusion in the study.
* Other pathologic conditions or circumstances that difficult participation in the study according to medical criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-12; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Safety evaluation | 24 weeks
  To determine the overall safety of RNL-JointStem® carrier using physical examinations, vital signs, treatment emergent adverse events (TEAEs), and the results of clinical lab tests.
WOMAC(Western Ontario and McMaster Universities) Index | 24 weeks
  Pain as measured by the The Western Ontario and McMaster Universities Arthritis Index (WOMAC) Pain Score.

SECONDARY OUTCOMES:
Magnetic Resonance Imaging | 24 weeks
  Changes in the MRI knee with cartilage mapping and clinical improvement assessed by radiologist.
KSCRS(Knee Society Clinical rating System) | 24 weeks
  Changes in exercise score and function of joint evaluation by KSCRS(Knee Society Clinical rating System).
VAS(11-point box visual analogue scale) | 24 weeks
  Changes in VAS(11-point box visual analogue scale) score.
Histological evaluates | 24 weeks
  Biopsy specimens subject to safranin-O staining and immunohistochemistry for type I and II collagen. Thickness of the articular cartilage before and after injection measure, and specimens evaluate with ICRS II by a blind histopathologist.

OTHER OUTCOMES:
cartilage volume of the knee joint | 24 weeks
  changes of the cartilage volume of the knee joint measure using a semi-automated segmentation method by a blinded researcher (webappendix)
Arthroscopy | 24 weeks
  Arthroscopy performs to evaluate any change in cartilage defect at the time of cell injection, and at 6 months after injection
X-ray | 24 weeks
  X-ray perform to measure with Kellgren-Lawrence grade,20 joint space width of the medial compartment,21 mechanical axis with weight bearing line,22 and anatomical axis.

CONTACTS AND LOCATIONS:
Overall Officials: Kang Sup Yoon, M.D. & Ph.D., Principal Investigator — SMG-SNU Boramae Hospital
Locations (1):
- SMG-SNU Boramae Hospital, Seoul, South Korea

REFERENCES:
- [Result] Jo CH, Lee YG, Shin WH, Kim H, Chai JW, Jeong EC, Kim JE, Shim H, Shin JS, Shin IS, Ra JC, Oh S, Yoon KS. Intra-articular injection of mesenchymal stem cells for the treatment of osteoarthritis of the knee: a proof-of-concept clinical trial. Stem Cells. 2014 May;32(5):1254-66. doi: 10.1002/stem.1634. PMID 24449146
- [Result] Jo CH, Chai JW, Jeong EC, Oh S, Shin JS, Shim H, Yoon KS. Intra-articular Injection of Mesenchymal Stem Cells for the Treatment of Osteoarthritis of the Knee: A 2-Year Follow-up Study. Am J Sports Med. 2017 Oct;45(12):2774-2783. doi: 10.1177/0363546517716641. Epub 2017 Jul 26. PMID 28746812